CLINICAL TRIAL: NCT07325006
Title: Impact of Physician Behavior on Cancer Distress
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ROR2503; NCI-2025-09164 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-011548 (Other: Mayo Clinic)
Record Dates: First submitted 2025-12-22; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete a survey and have their medical records reviewed on study. Patients who score a 7 or higher on the NCCN distress thermometer receive distress management patient education materials and recommendation to follow up with their care team.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This evaluates the impact of physician behaviors and other factors experienced during radiation treatment influence distress levels in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18+ years old)
* Must have a diagnosis of neoplasm
* Must be actively undergoing radiation therapy (RT) or have completed RT within the last month at Mayo Clinic in Rochester
* Able to read and write in English
* Must have email and Mayo Clinic patient portal access

Exclusion Criteria:

* Patients who have not yet started RT
* Patients who have been seen in consultation but not recommended for radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients who are undergoing or have completed radiation therapy within the last month at Mayo Clinic in Rochester
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Explore what physician behaviors contribute to patients' cancer distress | Baseline (at enrollment)
  Participants will indicate levels of distress on an 11-point Likert scale (10=extreme distress; 0=no distress). Physician behaviors that contribute to patients' cancer distress (as reported by patients) will be assessed using a free-text question. Topics and contextual factors will be identified by searching for themes with a thematic analysis. Descriptive statistics will be utilized to broadly analyze results. Data will initially be analyzed in its entirety. Subgroup analyses will then be done for patients who have vs have not experienced clinically significant distress (past or current score of 4+ on the distress thermometer). Additional subgroup analyses may be conducted depending on response.
Explore what physician behaviors lessen patients' cancer distress | Baseline (at enrollment)
  Participants will indicate levels of distress on an 11-point Likert scale (10=extreme distress; 0=no distress). Physician behaviors that lessen patients' cancer distress (as reported by patients) will be assessed using a free-text question. Topics and contextual factors will be identified by searching for themes with a thematic analysis. Descriptive statistics will be utilized to broadly analyze results. Data will initially be analyzed in its entirety. Subgroup analyses will then be done for patients who have vs have not experienced clinically significant distress (past or current score of 4+ on the distress thermometer). Additional subgroup analyses may be conducted depending on response.
Explore how non-physician factors in the patient care experience contribute to patients' cancer distress | Baseline (at enrollment)
  Participants will indicate levels of distress on an 11-point Likert scale (10=extreme distress; 0=no distress). Other factors that contribute to patients' cancer distress (as reported by patients) will be assessed using a free-text question. Topics and contextual factors will be identified by searching for themes with a thematic analysis. Descriptive statistics will be utilized to broadly analyze results. Data will initially be analyzed in its entirety. Subgroup analyses will then be done for patients who have vs have not experienced clinically significant distress (past or current score of 4+ on the distress thermometer). Additional subgroup analyses may be conducted depending on response.
Explore how non-physician factors in the patient care experience lessen patients' cancer distress | Baseline (at enrollment)
  Participants will indicate levels of distress on an 11-point Likert scale (10=extreme distress; 0=no distress). Other factors that lessen patients' cancer distress (as reported by patients) will be assessed using a free-text question. Topics and contextual factors will be identified by searching for themes with a thematic analysis. Descriptive statistics will be utilized to broadly analyze results. Data will initially be analyzed in its entirety. Subgroup analyses will then be done for patients who have vs have not experienced clinically significant distress (past or current score of 4+ on the distress thermometer). Additional subgroup analyses may be conducted depending on response.
Patient ratings of preference for physician-initiated conversations | Baseline (at enrollment)
  Patient ratings of preference for physician-initiated conversations on five sensitive topics: mental health, sexual health, financial health, cancer survival and mortality/prognosis, and personal relationship dynamics will be assessed using a study-specific survey. Responses are recorded on a Likert scale of 0-10 where 0=not at all and 10=very much so. Descriptive statistics will be utilized to analyze results.

CONTACTS AND LOCATIONS:
Overall Officials: May Elbanna, MB, BCh, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials